CLINICAL TRIAL: NCT01787955
Title: Impact of Braun Anastomosis on Reduction in Delayed Gastric Emptying Following Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2012-0879
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Periampullary Pathology Requiring Pancreaticoduodenectomy
Keywords: Pylorus preserving pancreaticoduodenectomy(PPPD), Delayed gastric emptying syndrome(DGE), Braun anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Braun anastomosis group (Experimental)
  Interventions: Procedure: PPPD with Braun anastomosis
- conventional group (Active Comparator): conventional Pylorus preserving pancreaticoduodenectomy
  Interventions: Procedure: conventional PPPD

INTERVENTIONS:
Procedure: PPPD with Braun anastomosis — making communication between E-loop and A-loop (Braun anastomosis 30cm away from duodenojejunostomy, by using staple method) will be added to conventional PPPD.
  Arms: Braun anastomosis group
Procedure: conventional PPPD
  Arms: conventional group

SUMMARY:
Pylorus preserving pancreaticoduodenectomy (PPPD) has been considered as only curative treatment modality for periampullary tumor. High mortality rates after PPPD have been reduced down to 1%. However, postoperative morbidities are still reported around 10 to 20 % even in high volume centers.The delayed gastric emptying syndrome(DGE) is one of major complications after PPPD. Many randomized control studies reported that pylorus preserving method was not related to the occurence of DGE. Thus,we assumed that large amount of biliary and pancreatic juice might affect DGE.

With the aim to prove that the use of Braun anastomosis after PPPD can prevent DGE, the investigators started the recruitment of patients with a periampullary tumors to this clinical trial from february 2013 with the study hypothesis that patients with Braun anastomosis had less DGE than those who only got conventional PPPD.

The investigators have calculated the number of patients necessaries to have statistical significant differences in 60 patients with a rate DGE expected to be higher than 30%.

The study include all the patients that usually arrive to our surgery department and who are indicated to PPPD for the curative treatment of periampullary tumor.

The study is randomized, double blind where the investigators and the patients do not know if the patients are in the Braun anastomosis group or not, and prospectively analyzed. All the clinical and laboratory or radiographic finds relative to the occurrence of DGE are recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with periampullary disease who have to be treated by PPPD

   * pancreatic cancer, distal bile duct cancer, duodenal cancer, and so on.
2. 20 year to 80 year-old patients
3. In terms of general performance status, the patients with more than 70% of the Karnofsky score or ECOG 0 to 1.

Exclusion Criteria:

1. Patients with unresectable or locally advanced and metastatic cancer.
2. The patient who does not want to take the operation.
3. The patient with more than 3 of ASA score.
4. Drug abusers or alcoholics.
5. Non-compliances
6. The patient who does not want to participate the clinical trials.
7. The patients who can not read or understand about informed consent form such as a mentally retarded person, the blind, illiteracy, or foreigner.
8. The patient who have previous transabdominal surgery
9. The patient who have to have resection of other organs or vessels other than standard PPPD
10. The patient who is indicated to laparoscopic PPPD

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Comparison of Delayed gastric emptying syndrome occurrence | 10 days after operation
  Comparison of DGE occurrence between Braun anastomosis group and conventional Pylorus preserving pancreaticoduodenectomy without Braun anastomosis group

CONTACTS AND LOCATIONS:
Locations (1):
- Severane hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Nikfarjam M, Houli N, Tufail F, Weinberg L, Muralidharan V, Christophi C. Reduction in delayed gastric emptying following non-pylorus preserving pancreaticoduodenectomy by addition of a Braun enteroenterostomy. JOP. 2012 Sep 10;13(5):488-96. doi: 10.6092/1590-8577/800. PMID 22964955